CLINICAL TRIAL: NCT04705246
Title: Effect of Psychoeducation Upon Exposure to Sounds and Hyperacusis Severity
Brief Title: Role of Exposure in Hyperacusis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exposure in Hyperacusis
Record Dates: First submitted 2020-11-04; First posted 2021-01-12 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Hyperacusis
MeSH Terms: conditions — Hyperacusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psychoeducation (Experimental): The goal of the psychoeducation session is to provide insight in the hyperacusis symptoms, take away the fear of external noises, and encourage exposure to noise.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — The goal of the psychoeducation session is to provide insight in the hyperacusis symptoms, take away the fear of external noises, and encourage exposure to noise.

SUMMARY:
This study focuses on patients with a primary complaint of hyperacusis. Hyperacusis has been defined as 'abnormally reduced tolerance to sound'. It shows a high comorbidity with tinnitus, the perception of sound in the absence of a sound source. For the period of one month, hyperacusis and tinnitus severity and exposure to sounds will be evaluated by use of Ecological Momentary Assessment (EMA) in all participants. A novel approach to assessments, EMA prompts participants during their daily life to answer short questionnaires, increasing ecological validity and minimizing the risk for recall and memory biases. At a randomized time point during the one-month period, participants will individually receive a single psychoeducation session (1h) delivered by an experienced audiologist. The goal of the study is to investigate if the psychoeducation session leads to an increase in exposure to sound and a decrease in hyperacusis severity.

ELIGIBILITY:
Inclusion Criteria:

* primary complaint of hyperacusis

Exclusion Criteria:

* primary complaint of misophonia
* primary complaint of tinnitus
* undergoing another therapy at the moment of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in EMA questions from baseline to end of the study | 8 random time points each day during the period of the study, from baseline and after intervention, though study completion for an average of 1 month
  Change in questions concerning exposure, hyperacusis and tinnitus during the day from baseline measurement to last day of the study period

SECONDARY OUTCOMES:
Hyperacusis Questionnaire | before intervention, immediately post intervention
  Hyperacusis severity self-report questionnaire, ranging from 0-42 with a higher score representing a higher sensitivity to sounds. A score of 28 is the cut-off for auditory hypersensitivity.
Tinnitus Functional Index (TFI) | before intervention, immediately post intervention
  Tinnitus severity self-report questionnaire, ranging from 0-100 with a higher score representing a more severe tinnitus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blaesing L, Kroener-Herwig B. Self-reported and behavioral sound avoidance in tinnitus and hyperacusis subjects, and association with anxiety ratings. Int J Audiol. 2012 Aug;51(8):611-7. doi: 10.3109/14992027.2012.664290. Epub 2012 Mar 24. PMID 22443320
- [Background] Goldberg RL, Piccirillo ML, Nicklaus J, Skillington A, Lenze E, Rodebaugh TL, Kallogjeri D, Piccirillo JF. Evaluation of Ecological Momentary Assessment for Tinnitus Severity. JAMA Otolaryngol Head Neck Surg. 2017 Jul 1;143(7):700-706. doi: 10.1001/jamaoto.2017.0020. PMID 28448659
- [Background] Henry JA, Thielman E, Zaugg T, Kaelin C, Choma C, Chang B, Hahn S, Fuller B. Development and field testing of a smartphone "App" for tinnitus management. Int J Audiol. 2017 Oct;56(10):784-792. doi: 10.1080/14992027.2017.1338762. Epub 2017 Jul 2. PMID 28669224
- [Background] Kratochwill TR, Levin JR. Enhancing the scientific credibility of single-case intervention research: randomization to the rescue. Psychol Methods. 2010 Jun;15(2):124-44. doi: 10.1037/a0017736. PMID 20515235